CLINICAL TRIAL: NCT04416776
Title: Validation of the Utility of Strabismus Intelligent Diagnostic System: A Clinical Trial
Brief Title: Validation of the Utility of Strabismus Intelligent Diagnostic System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: SIDS-2020
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Ophthalmological Disorder; Strabismus
MeSH Terms: conditions — Eye Diseases; Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eligible patients for AI test: Device: strabismus diagnostic system.
  Interventions: Drug: Strabismus diagnostic system.

INTERVENTIONS:
Drug: Strabismus diagnostic system. — An AI platform based on corneal light-reflection photos to facilitate the diagnosis and angle evaluation of strabismus and to provide advice for surgical planning.

SUMMARY:
Strabismus affects approximately 0.8%-6.8% of the world's population and appears by the age of 3 years in 65% of affected individuals. Manual measurement of deviation is often laborious and highly dependent on the experience of the specialist and the cooperation of the patients. Current strabismus evaluation technologies are heavily dependent on model eyes. Here, the investigators use deep learning to develop an artificial intelligence (AI) platform consisting of three deep learning (DL) systems to screen strabismus, evaluate deviation and propose a surgical plan based on corneal light-reflection photos. The investigator also conduct clinical trial to validate its versatility in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the outpatient clinic of strabismus department.

Exclusion Criteria:

* Patients or their parents diagree to participate in the trial.
* Patients with blepharoptosis.
* Patients can't facing forward or lacking fixation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A prospective study to validate the accuracy of the strabismus intelligent diagnostic system in the clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of accurate, mistaken and miss detection of the diagnostic system. | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China